CLINICAL TRIAL: NCT04266093
Title: Gene Therapy Follow up Protocol for Subjects Previously Enrolled in NCI Center for Immuno-Oncology Studies
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 200051; 20-C-0051
Record Dates: First submitted 2020-02-11; First posted 2020-02-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-30

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Neoplasms; Oropharyngeal Neoplasms; Squamous Intraepithelial Lesions of the Cervix; Hematologic Malignacies
Keywords: Gene Transfer; Recombinant DNA Product; Gamma-Retroviral Vectors; Laboratory Evaluation; Natural History
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Oropharyngeal Neoplasms; Squamous Intraepithelial Lesions of the Cervix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects who have enrolled on an applicable NCI CIO gene therapy treatment protocol.
  Interventions: Drug: GeneTherapy

INTERVENTIONS:
Drug: GeneTherapy — Observation/ Gene Therapy Long-term Follow-up. Subjects who have enrolled on an applicable NCI CIO gene therapy treatment protocol.

SUMMARY:
Background:

Gene therapy is closely followed by the U.S. Food and Drug Administration (FDA). The FDA requires researchers to conduct long-term follow-up of people who have had the treatment. This study collects data on people who have had gene therapy and sends it to the FDA. The data does not include participants names.

Objective:

To contact current or past participants of gene therapy protocols at least once a year for up to 15 years to ensure they have not had any harmful side effects.

Eligibility:

People aged 18 and older who have had gene therapy in a National Cancer Institute study

Design:

Participants will give their address and telephone number. They will also give and the address and phone number of 1 or 2 other people who will know where they are.

For the first year after gene therapy, participants will give blood samples 3 times (at 3, 6, and 12 months). For the next 4 years, they may have a physical exam and laboratory tests with a home physician. They will get a kit to mail in blood samples. Or they can visit the NIH Clinical Center. They will be asked if they have had any signs of neurological, autoimmune, or blood disorders, or any new cancers.

For years 6 to 15, participants will be contacted yearly via phone or email and asked questions about their health. They may give blood samples.

When the participant dies, if researchers think the death was caused by gene therapy, they will ask the participant s family to allow an autopsy.

DETAILED DESCRIPTION:
Background:

The NCI CIO conducts clinical trials utilizing gene transfer. The current FDA requirements for long term follow up may be up to fifteen years for some products. As this time period is frequently longer than studies are expected to be open, a protocol is necessary to ensure the necessary follow up of these subjects

Objectives:

To facilitate collection of long term follow up information on subjects who have participated in gene transfer studies as required by the U.S. Food and Drug Administration and other regulatory groups

Eligibility:

Enrollment on a NCI CIO treatment protocol for gene therapy.

Design:

Patients will undergo physical exams, laboratory evaluations and/or phone follow up as required by the treatment protocol and/or as clinically indicated.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects who have enrolled on an applicable NCI CIO gene therapy treatment protocol. Age >= 18 years. Note: Children are generally excluded from CIO gene therapy studies and inclusion on this follow-up study will be limited to 18 years and older.

EXCLUSION CRITERIA:

-Children

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To facilitate collection of long term follow up information on subjects who have participated in gene transfer studies as required by the U.S. Food and Drug Administration and other regulatory groups
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-08 (Actual); Primary Completion 2035-10-01 (Estimated); Study Completion 2050-10-01 (Estimated)

PRIMARY OUTCOMES:
To provide long term follow up of patients previously enrolled on treatment protocols in the NCI CIO. | 15 years
  List of long time adverse event frequency after Gene therapy drug

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Norberg, D.O., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0051.html